CLINICAL TRIAL: NCT04958369
Title: Comparison of the Ultrasound-guided Axillary Vein Puncture With the Conventional Cephalic Vein Cut-down Technique for Implantation of Cardiac Devices
Brief Title: Ultrasound-guided Axillary Versus Conventional Cephalic Venous Access for Implantation of Cardiac Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Georgios Leventopoulos, Consultant Cardiologist, University Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 93/01.03.2021
Record Dates: First submitted 2021-06-27; First posted 2021-07-12 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Pacemaker; Implantable Cardioverter-defibrillator
Keywords: pacemaker; implantable cardioverter-defibrillator; axillary vein; cephalic vein; ulatraound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided axillary venous access (Active Comparator): Cardiac device implantation will be performed with ultrasound-guided axillary venous access.
  Interventions: Device: Ultrasound-guided axillary venous access
- Cephalic venous access (Active Comparator): Cardiac device implantation will be performed with conventional cephalic venous access (cut-down technique).
  Interventions: Device: Cephalic venous access

INTERVENTIONS:
Device: Ultrasound-guided axillary venous access — Venous access is obtained through ultrasound-guided axillary vein puncture and Seldinger technique.
  Arms: Ultrasound-guided axillary venous access
Device: Cephalic venous access — Venous access is obtained through cephalic vein cut-down.
  Arms: Cephalic venous access

SUMMARY:
The implantation of cardiac electronic devices is a common procedure in the Electrophysiology Laboratory. The most commonly used venous access sites are the cephalic, the axillary and the subclavian vein.

Studies comparing these options have been conducted in the past. Axillary venous access can be achieved either through axillary vein angiography or by ultrasound guidance. Nevertheless, appropriate training is required for the ultrasound-guided axillary puncture technique-as well as for the cephalic vein cutdown technique.

Data from randomized trials regarding direct comparison of the two methods in terms of efficacy and safety are very limited.

The purpose of the study is the comparison of the efficacy and safety of the ultrasound-guided axillary venous access technique versus the cephalic venous access using the cut-down technique in patients requiring intravenous cardiac device (single-chamber/dual-chamber pacemaker/defibrillator) implantation.

DETAILED DESCRIPTION:
This study is a single-center, randomized, clinical trial. Its purpose is the comparison of the ultrasound-guided axillary venous access technique versus the cephalic venous access using the cut-down technique in cardiac device implantation procedures. Prerequisite for starting patients' recruitment is that the operators have undergone a training phase in ultrasound-guided axillary vein puncture in the Interventional Radiology Laboratory and have completed at least 30 procedures. A GE V-scan device with a special linear transducer for vessel examination will be utilized for the ultrasound guidance. Micropuncture technique will be performed for venous access.

Eligibility criteria:

Inclusion criteria

* Age ≥ 18 years
* Indication for single- or dual-chamber pacemaker of defibrillator implantation
* Written informed consent Exclusion criteria
* Indication for biventricular pacemaker or defibrillator
* Upgrade in pacing or defibrillation system

After the operators' training phase, candidates for pacemaker or defibrillator (single- or dual-chamber) implantation who fulfill the inclusion criteria will be randomly assigned with 1:1 allocation to one of the Groups:

A. ultrasound-guided axillary venous access B. cephalic venous access through the cut-down technique In case of access failure in Group A, the alternative puncture options are through the cephalic vein, the axillary vein with angiography guidance, the axillary vein without angiography guidance or the subclavian vein. In case of access failure in Group B which includes the insertion of only one lead wire or none, the alternative puncture options are through the axillary vein with angiography, the axillary vein without angiopraghy or the subclavian vein.

Data of the study participants that will be recorded include: demographics, Body Mass Index (BMI), cardiovascular risk factors, comorbidities, indication for cardiac device implantation, type of device (pacemaker/defibrillator, single-chamber/dual-chamber), side of implantation (right, left), type of pocket (subcutaneous, submuscular).

Regarding NOAC administration, patients will undergo the implantation procedure after cessation of rivaroxaban for at least 20 hours before the procedure and apixaban or dabigatran for at least 16 hours before the procedure. Longer periods of cessation will be applied in patients with renal dysfunction. In patients on treatment with acenocoumarol or warfarin, procedures will be performed without discontinuation of the drugs with target INR=2.

Regarding anticoagulation management in patients with mechanical valves the following anticoagulation management plan will be applied: i) in patients with metallic aortic valve, no discontinuation of anticoagulation with target INR=2 and ii) in patients with metallic mitral valve, no discontinuation of anticoagulation, with target INR<3-4.

The study hypothesis is that ultrasound-guided axillary venous access will lead to a higher rate of successful implantation procedures compared to cephalic vein access through the cut-down technique.

Based on available research data and pilot data, the hypothesis is that the success rate in ultrasound-guided axillary venous access group will be 90% compared to 65% in the cephalic venous access group. A sample size of 57 patients in each group is expected to offer statistic power of 90% (a=0.05, two-tailed) to the aforementioned result.

The study has been approved by the Ethics Committee of the University Hospital of Patras. All candidates will participate after written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Indication for single- or dual-chamber pacemaker of defibrillator implantation
* Written informed consent

Exclusion Criteria:

* Indication for biventricular pacemaker/defibrillator
* Upgrade in pacing or defibrillation system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Rate of successful cardiac device implantation | Intervention time (Day 0)

SECONDARY OUTCOMES:
Duration of lead insertion procedure | Intervention time (Day 0)
  Time from the administration of local anesthesia to the insertion of leads into the inferior vena cava
Total procedure duration | Intervention time (Day 0)
  Time from the administration of local anesthesia to skin suture
Radiation dose | Intervention time (Day 0)
Fluoroscopy time | Intervention time (Day 0)
Procedure-related complication rate (pneumothorax, cardiac tamponade, pocket hematoma, lead displacement, fever, need for antibiotic treatment) | Day 0-30
  All procedure related complications including pneumothorax, cardiac tamponade, pocket hematoma, lead displacement, fever, need for antibiotic treatment
Pain associated with the procedure assessed by use of the visual analogue pain scale from 0 to 10 (0: no pain, 10: worse pain) | Day 1
  Pain associated with the procedure assessed by use of the visual analogue pain scale from 0 to 10 (0: no pain, 10: worse pain)
Duration of hospitalization | Through study completion, an average of 1.5 year
  The number of days from the day of implantation till the day of hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Patras, Pátrai, Rion, Greece

IPD SHARING:
Plan to Share IPD: No